CLINICAL TRIAL: NCT05285826
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Clinical Study to Evaluate the Efficacy, Immunogenicity, and Safety of V503, a 9-Valent Human Papillomavirus (HPV) Vaccine, in Chinese Males 20 to 45 Years of Age
Brief Title: Efficacy, Immunogenicity, and Safety of V503 in Chinese Males (V503-052)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V503-052
Record Dates: First submitted 2022-03-08; First posted 2022-03-18 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Papillomavirus Infections
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- V503 (Experimental): Participants will receive a single 0.5 mL intramuscular (IM) injection of V503 at Day 1, Month 2, and Month 6.
  Interventions: Biological: 9vHPV Vaccine
- Placebo (Placebo Comparator): Participants will receive a single 0.5 mL IM injection of placebo at Day 1, Month 2, and Month 6.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: 9vHPV Vaccine — 9-valent human papillomavirus (Types 6, 11, 16, 18, 31, 33, 45, 52, 58) L1 virus-like particle vaccine administered as a 0.5-mL IM injection
  Other Names: V503
  Arms: V503
Other: Placebo — Sterile saline solution administered as a 0.5 mL IM injection
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy, immunogenicity, and safety of 9-valent human papillomavirus (9vHPV; V503) vaccine in Chinese men 20 to 45 years of age. It will enroll heterosexual men (HM) and men who have sex with men (MSM), will be stratified by age and sexual orientation, and will have two stages. The primary hypothesis of Stage I is: 9vHPV vaccine reduces the combined incidence of HPV 6-, 11-, 16-, 18-, 31-, 33-, 45-, 52-, and 58-related external genital and intra-anal 12-month persistent infection (PI) compared with placebo in males 20 to 45 years of age who are seronegative at Day 1 and polymerase chain reaction (PCR) negative from Day 1 through one month post-Dose 3 to the relevant HPV type. The primary hypothesis of Stages I and II combined is: 9vHPV vaccine reduces the combined incidence of HPV 6-, 11-, 16-, 18-, 31-, 33-, 45-, 52-, and 58-related genital warts, penile/perianal/perineal intraepithelial neoplasia (PIN), or penile/perianal/perineal cancer compared with placebo in males 20 to 45 years of age who are seronegative at Day 1 and PCR negative from Day 1 through one month post-Dose 3 to the relevant HPV type.

ELIGIBILITY:
Inclusion Criteria:

* Is a Chinese male.
* Has no more than 5 lifetime sexual partners.

Exclusion Criteria:

* Has a history of known prior vaccination with an HPV vaccine.
* Has a history of HPV-related external genital lesions, HPV-related intra-anal lesions, or HPV-related head and neck cancer.
* Has a history of severe allergic reaction that required medical intervention.
* Has received immune globulin or blood-derived products in the past 3 months or plans to receive any before Month 7 of the study.
* Has a history of splenectomy, is currently immunocompromised, or has been diagnosed with immunodeficiency, human immunodeficiency virus (HIV), lymphoma, leukemia, systemic lupus erythematosus, rheumatoid arthritis, juvenile rheumatoid arthritis, inflammatory bowel disease, or other autoimmune condition.
* Has received immunosuppressive therapy in the past year, excluding inhaled, nasal, or topical corticosteroids and certain regimens of systemic corticosteroids.
* Has a known thrombocytopenia or coagulation disorder that would contraindicate IM injections.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8100 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2029-05-25 (Estimated); Study Completion 2029-05-25 (Estimated)

PRIMARY OUTCOMES:
Stage I: Combined Incidence of HPV 6-, 11-, 16-, 18-, 31-, 33-, 45-, 52-, and 58-related External Genital and Intra-anal 12-month Persistent Infection | Up to approximately 30 months
  This endpoint is defined as having occurred if a participant is positive for the same HPV type by the HPV PCR assay in the penile, scrotum, perineal, perianal and intra-anal swabs, biopsy, or excised samples obtained in 3 or more consecutive visits over a period of at least 12 months.
Stages I and II: Combined Incidence of HPV 6-, 11-, 16-, 18-, 31-, 33-, 45-, 52-, and 58-related Genital Warts, PIN, or Penile/Perianal/Perineal Cancer | Up to approximately 78 months
  This endpoint is defined as having occurred if on a single biopsy or excised tissue from a participant, there is: (a) a pathology panel consensus diagnosis of genital warts, PIN of any grade, or penile/perianal/perineal cancer; and (b) detection of at least 1 of HPV types 6, 11, 16, 18, 31, 33, 45, 52 or 58 by Thinsection PCR in an adjacent section from the same tissue block.

SECONDARY OUTCOMES:
Stage 1: Combined Incidence of HPV 6-, 11-, 16-, 18-, 31-, 33-, 45-, 52-, and 58-related External Genital and Intra-anal 6-month Persistent Infection | Up to approximately 30 months
  This endpoint is defined as having occurred if a participant is positive for the same HPV type by the HPV PCR assay in the penile, scrotum, perineal, perianal and intra-anal swabs, biopsy, or excised samples obtained in 2 or more consecutive visits over a period of at least 6 months.
Stage 1: Geometric Mean Titers (GMTs) to HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 at One Month Post-Dose 3 | Month 7
  GMTs to HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 will be measured with a Competitive Luminex Immunoassay (cLIA).
Stage 1: Percentage of Participants Achieving Seroconversion to HPV 6, 11, 16, 18, 31, 33, 45, 52, or 58 at One Month Post-Dose 3 | Month 7
  A participant who changes serostatus from seronegative at Day 1 to seropositive at one month post-Dose 3 for a given HPV type is considered to have achieved seroconversion for that type. A participant with a titer at or above the seropositivity cutoff for a given HPV type, as measured by cLIA, is considered seropositive for that type.
Stage I: Percentage of Participants Who Report at Least 1 Solicited Injection-site Adverse Event (AE) | Day 1 through Day 8 following any vaccination
  An AE is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study vaccine. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or a protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the study vaccine or protocol-specified procedure is also an AE. Solicited injection-site AEs such as erythema, swelling, pain, and induration at the injection site will be recorded.
Stage I: Percentage of Participants Who Report at Least 1 Solicited Systemic AE | Day 1 through Day 8 following any vaccination
  An AE is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study vaccine. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or a protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the study vaccine or protocol-specified procedure is also an AE. Systemic AEs are those not categorized as injection-site AEs.
Stage I: Percentage of Participants Who Experience at Least 1 Serious Adverse Event (SAE) | Up to approximately 30 months
  An AE is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study vaccine. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or a protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the study vaccine or protocol-specified procedure is also an AE. An SAE is an AE that results in death, is life threatening, results in a persistent or significant disability or incapacity, results in or prolongs an existing hospitalization, is a congenital anomaly or birth defect, or is another important medical event.
Stages I and II: Combined Incidence of HPV 6-, 11-, 16-, 18-, 31-, 33-, 45-, 52-, and 58-related Anal Intraepithelial Neoplasia (AIN) or Anal Cancer (MSM participants only) | Up to approximately 78 months
  This endpoint is defined to have occurred if on a single biopsy or excised tissue from a participant, there is: (a) a pathology panel consensus diagnosis of AIN of any grade or anal cancer; and (b) detection of at least 1 of HPV types 6, 11, 16, 18, 31, 33, 45, 52 or 58 by Thinsection PCR in an adjacent section from the same tissue block.
Stages I and II: Percentage of Participants Who Experience at Least 1 SAE | Up to approximately 78 months
  An AE is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study vaccine. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or a protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the study vaccine or protocol-specified procedure is also an AE. An SAE is an AE that results in death, is life threatening, results in a persistent or significant disability or incapacity, results in or prolongs an existing hospitalization, is a congenital anomaly or birth defect, or is another important medical event.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (34):
- China (34):
  - Beijing Youan Hospital ( Site 0001), Beijing, Beijing Municipality
  - The Second Affiliated Hospital Chongqing Medical University ( Site 0052), Chongqing, Chongqing Municipality
  - Chongqing Public Health Medical Center ( Site 0003), Chongqing, Chongqing Municipality
  - The First Hospital of Lanzhou University ( Site 0034), Lanzhou, Gansu
  - Southern Medical University Nanfang Hospital-Center for Drug Clinical Research ( Site 0031), Guangzhou, Guangdong
  - The University of Hong Kong - Shenzhen Hospital ( Site 0049), Shenzhen, Guangdong
  - Center for Disease Control and Prevention of Rong An ( Site 0046), Liuchow, Guangxi
  - Liucheng County Centers for Disease Control and Prevention ( Site 0045), Liuchow, Guangxi
  - Wuhan Union Hospital ( Site 0032), Wuhan, Hubei
  - Hunan Provincial Center for Disease Control and Prevention ( Site 0040), Changsha, Hunan
  - The Third Xiangya Hospital of Central South University ( Site 0033), Changsha, Hunan
  - Loudi Disease Prevention and Control Center Zhiyebing Prevention And Treatment Hospital ( Site 0015), Louxing District, Hunan
  - Xiangtan Disease Prevention and Control Center ( Site 0030), Xiangtan, Hunan
  - Xiangxiang Disease Prevention and Control Center ( Site 0016), Xiangxiang, Hunan
  - Qiyang Center for Disease Control and Prevention ( Site 0014), Yongzhou, Hunan
  - The Second Hospital of Nanjing (Tangshan Branch) ( Site 0028), Nanjing, Jiangsu
  - The first affiliated hospital of China medical university ( Site 0041), Shenyang, Liaoning
  - Liaoning University of Traditional Chinese Medicine Affiliated Hospital ( Site 0048), Shenyang, Liaoning
  - Yuanqu Center for Disease Control and Prevention ( Site 0019), Yuncheng, Shanxi
  - Yanhu Center for Disease Control and Prevention of Yuncheng ( Site 0018), Yuncheng, Shanxi
  - Yongji Center for Disease Control and Prevention ( Site 0026), Yuncheng, Shanxi
  - Ruicheng Center for Disease Control and Prevention ( Site 0025), Yuncheng, Shanxi
  - Dazhu Disease Prevention and Control Center ( Site 0010), Dazhou, Sichuan
  - Yuechi Disease Prevention and Control Center ( Site 0009), Guang’an, Sichuan
  - Mianyang Center for Disease Control and Prevention ( Site 0007), Mianyang, Sichuan
  - Santai County Center for Disease Control and Prevention ( Site 0008), Mianyang, Sichuan
  - Neijiang Center for Disease Control and Prevention ( Site 0011), Neijiang, Sichuan
  - Tianjin Second People's Hospital ( Site 0004), Tianjin, Tianjin Municipality
  - Tianjin People' s Hospital ( Site 0038), Tianjin, Tianjin Municipality
  - Binchuan County Center for Disease Control and Prevention ( Site 0022), Dali, Yunnan
  - Xiangyun County Center for Disease Control and Prevention ( Site 0021), Dali, Yunnan
  - First Affiliated Hospital of Kunming Medical University ( Site 0051), Kunming, Yunnan
  - Yunnan Provincial Infectious Disease Hospital ( Site 0042), Kunming, Yunnan
  - Zhejiang University School of Medicine - Affiliated Wenzhou Traditional Chinese Medicine Hospital (W, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/